CLINICAL TRIAL: NCT01966809
Title: A Phase II Study of Photodynamic Therapy (PDT) With Photofrin® (IND 104,613) For Recurrent High Grade Gliomas in Adults
Brief Title: Photodynamic Therapy (PDT) For Recurrent High Grade Gliomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment.
Sponsor: Harry T Whelan, MD (Other)
Collaborators: Pinnacle Biologics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Harry T Whelan, MD, Bleser Professor of Neurology, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00023580
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Brain Tumor, Recurrent
Keywords: Brain Tumor; Photodynamic Therapy; Photochemotherapy; Astrocytoma; Pilocytic Astrocytoma; Low grade Astrocytoma; Anaplastic Astrocytoma; Glioblastoma; GBM; Chordoma; Germinoma; Germ Cell Tumor; Non-germinoma; CNS Lymphoma; Craniopharyngioma; Mixed Glioma; Optic Nerve Glioma; Meningioma; Oligodendroglioma; Pituitary Tumors; Desmoplastic Neuroepithelial Tumor; DNET; glioblastoma multiforme; glioma; glioblastoma survivors; what is glioblastoma; gbm cancer; oligoastrocytoma; gbm tumor; anaplastic oligodendroglioma; High-Grade Glioma; high grade glioma; glioblastomas; glioblastoma cancer; anaplastic oligoastrocytoma; astrocytoma glioma; glioblastoma clinical trials; photodynamic therapy for cancer; glioblastoma multiforme clinical trials; astrocytoma glioblastoma; gbm grade 4; clinical trials for glioblastoma; photodynamic therapy cancer; clinical trials glioblastoma; glioblastoma clinical trials 2015; glioblastoma clinical trials 2014 not open in 2014; glioblastoma trials; gbm clinical trials; glioblastoma immunotherapy; malignant gliomas; anaplastic astrocytomas; immunotherapy for glioblastoma; immunotherapy glioblastoma; High Grade Glioblastoma Multiforme; clinical trial glioblastoma; glioblastoma clinical trial; glioblastoma trial; brain tumors; recurrent brain tumors; glioma grade 3; grade 3 brain tumor; grade 4 brain tumor
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma; Glioblastoma; Chordoma; Germinoma; Neoplasms, Germ Cell and Embryonal; Craniopharyngioma; Glioma; Optic Nerve Glioma; Meningioma; Oligodendroglioma; Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Photofrin photodynamic therapy. (Experimental): Photofrin photodynamic therapy. Drug - 2.5 mg/kg, light - 240 mJ/cm2.
  Interventions: Drug: Photofrin photodynamic therapy.

INTERVENTIONS:
Drug: Photofrin photodynamic therapy. — The subjects will receive a dose of 2.5 mg/kg of Photofrin intravenously 24 hours before planned surgical resection. Tumor resection will be carried out in the standard fashion in order to achieve the maximum tumor resection compatible with preservation of neurological function. After resection, Intralipid will be infused into the craniotomy and kept for approximately 45 min, while PDT will be performed. The illumination time will be calculated from the power density (mW) emitted by the laser and the radius (r) of the cavity to deliver a total light dose of 240 J/cm2 at a using the following formula:
  Treatment Time (sec) = Light dose (J/cm2) x Cavity surface (cm2) x 1000 Power density (mW) Cavity Surface (cm2) = 4 x 3.14 x r2 The optical fiber will be placed in the center of the surgical cavity and photoillumination will commence. After PDT, the Intralipid solution will be removed and the wound will be closed. The subject will be sent to the intensive care area for recovery.

SUMMARY:
This study will be aimed at investigating the effectiveness of a treatment for brain tumors called Photodynamic Therapy, or PDT. Briefly, a subject will receive a light-sensitive drug, called Photofrin®, the day before a tumor removal surgery. The next day, after the tumor is removed, red light from a laser will be shone into the tumor cavity through a light-diffusing sphere. This light will activate the photosensitizer, and possibly kill any tumor cells that may be left.

We plan to measure how long the subject may go without a new tumor regrowth, and overall how long subjects survive. We will compare these results to typical results to see if we are seeing any improvements.

Objective: To define the antitumor activity of Photofrin® and laser light activation within the confines of a Phase II study.

DETAILED DESCRIPTION:
Photodynamic therapy (PDT) is a well-known treatment for other type of tumors; however it is an experimental treatment for brain tumors. There is much we do not know about the effectiveness of PDT in patients with brain tumors. The purpose of this study is to define the antitumor activity of Photofrin® and laser light activation. Photofrin® is a photosensitizing drug (a dye that is activated by light) used in PDT. We want to test the activity of PDT and to see what are the effects (good and bad) on you and your brain tumor. We also want to learn if this treatment will cause brain tumors to shrink and whether it will help patients with brain tumors to live longer.

PDT is a cancer treatment that involves giving a photosensitive dye (Photofrin®), into your vein through a tube (called an IV). This dye will go inside of the cancer cells more than it will go inside the normal, healthy cells. PDT using Photofrin® is an approved treatment in patients with certain types of cancer such as lung, and esophageal (from the mouth to the stomach) cancers.

Everyone in this study will receive Photofrin® (porfimer sodium) for injection (Pinnacle Biologics, Inc., Bannockburn, IL, USA), and be treated with red light emitted by a red laser. The light will be sent from the laser to the surface of the brain where the tumor is located using a light transmitting fiber. The fiber will have a knob at the end that spreads the light out evenly in all directions.

Previous studies have shown that patients with malignant brain tumors called gliomas had a good response to PDT. The patients in these studies lived longer than they were expected to live. In one study of adults with brain tumors in Australia, patients given PDT had greatly improved survival rates. Fifty seven percent (57%) of the patients with gliomas called anaplastic astrocytoma survived for 36 months. Thirty seven percent (37%) of the patients with gliomas called glioblastoma multiforme survived for 36 months. Froedtert Hospital, in Milwaukee WI, has been involved in PDT studies in adults in the past. This current study is is being done in a very similar way to the study done in Australia, and will use increased Photofrin®) and light doses than our previous study.

ELIGIBILITY:
Inclusion Criteria

1. Age: Greater than or equal to 18 years of age.
2. Disease: Patients with relapsed or refractory high grade glioma are eligible. Patients must have had histologic verification of malignancy at original diagnosis or relapse. Tumors must be supratentorial in location.
3. Disease Status: Patients must have potentially resectable disease.
4. Therapeutic Options: Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
5. Performance Level: Karnofsky 50% or greater. Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
6. Predictable Life Expectancy: > 8weeks
7. Prior Therapy: Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy. At least three weeks from previous chemotherapy and 4 weeks from prior radiation therapy.
8. Organ Function:

   a. Adequate bone marrow function i. Absolute neutrophil count ≥ 1,000 ii. Platelet count ≥ 100,000 (may transfuse to meet requirement) b. Adequate renal function i. Creatinine clearance or radioisotope GFR ≥ 60 mL/min/1.73 m2 or ii. A serum creatinine within normal range based on age/gender. c. Adequate liver function i. Bilirubin (direct) ≤ 3X upper limit of normal (ULN) for age ii. SGPT (ALT) ≤ 10X ULN. For the purpose of this study, the ULN for SGPT is 45 U/L.

   iii. Serum albumin ≥ 2 g/dL. d. Adequate coagulation i. PT and INR ≤ 2X ULN for age.
9. Central Nervous System Function: Patients with seizure disorder may be enrolled if receiving non-enzyme inducing anticonvulsants and well controlled.
10. Informed Consent: All patients or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
11. Archival tumor tissue slides from initial diagnosis should be reviewed by Froedtert Health-MCW neuropathologist prior to study enrollment whenever possible.

Exclusion Criteria

1. Disseminated disease
2. Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study, as risks of fetal and teratogenic adverse effects of Photofrin® are not known.
3. Other concurrent tumor therapy
4. Subjects with porphyria
5. Subjects taking potentially photosensitizing drugs (Appendix 3)
6. The presence of adverse events of neurologic function, photosensitivity, or photophobia Grade 4 or higher (CTCAE Version 4.02).47
7. Allergy to eggs, soybean oil, or safflower oil (due to potential allergy against intralipids)
8. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-06; Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry T Whelan, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/ Froedtert Hospital, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Photofrin Photodynamic Therapy.: Photofrin photodynamic therapy. Drug - 2.5 mg/kg, light - 240 mJ/cm2.
  Photofrin photodynamic therapy.: The subjects will receive a dose of 2.5 mg/kg of Photofrin intravenously 24 hours before planned surgical resection. Tumor resection will be carried out in the standard fashion in order to achieve the maximum tumor resection compatible with preservation of neurological function. After resection, Intralipid will be infused into the craniotomy and kept for approximately 45 min, while PDT will be performed. The illumination time will be calculated from the power density (mW) emitted by the laser and the radius (r) of the cavity to deliver a total light dose of 240 J/cm2 at a using the following formula:
  Treatment Time (sec) = Light dose (J/cm2) x Cavity surface (cm2) x 1000 Power density (mW) Cavity Surface (cm2) = 4 x 3.14 x r2 The optical fiber will be placed in the center of the surgical cavity and photoillumination will commence.
Period: Overall Study
Arm/Group | Photofrin Photodynamic Therapy.
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Photofrin Photodynamic Therapy.
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Six Month Relapse-free Survival (RFS).
Description: Relapse free survival is the proportion of subjects who have gone six months since PDT without the disease getting worse.
Time Frame: Six months from PDT
Measure: Number; unit: participants
Arm/Group | Photofrin Photodynamic Therapy.
Number analyzed (Participants) | 1
participants | 0

2. Secondary Outcome: Remission Rate.
Description: To obtain preliminary data toward determining whether this combination results in higher remission rate when compared to historical data.
Time Frame: Three years from PDT
Population: Study closed before three year period was completed. Only one participant was enrolled.
Arm/Group | Photofrin Photodynamic Therapy.
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival and Overall Survival.
Description: To further explore and report progression-free survival and overall survival for three years post PDT treatment.
Time Frame: Three years from PDT
Population: Study closed before three year period was completed. Only one participant was enrolled.
Arm/Group | Photofrin Photodynamic Therapy.
Number analyzed (Participants) | 0

4. Secondary Outcome: Tumor Response.
Description: To measure complete response, partial response, stable disease or progressive disease using the response assessment for Neuro-Oncology (RANO) criteria with the follow-up medical imaging, which specifically incorporates volumetric measurements of brain tumor enhancement and clinical measures of neurological decline and to compare these outcomes to historical controls.
Time Frame: Six months from PDT
Population: Participant lost to followup before secondary outcome was assessed.
Arm/Group | Photofrin Photodynamic Therapy.
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Photofrin Photodynamic Therapy.
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photofrin Photodynamic Therapy. (N=1)
Altered mental status (Nervous system disorders) | 1 (1) — Change in the patient's mentation as well as decreased strength on the right side.

LIMITATIONS AND CAVEATS:
Early termination with only one participant enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT01966809/Prot_SAP_000.pdf